CLINICAL TRIAL: NCT04627103
Title: A Trial for a Procedure for Duodenal-Ileal Diversion With a Sleeve Gastrectomy for Patients With Obesity and Type 2 Diabetes Mellitus
Brief Title: Procedure for Duodenal-Ileal Diversion With a Sleeve Gastrectomy for Patients With Obesity and Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIW 20-001
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Obesity; Diabetes Mellitus; Diabetes Mellitus, Type 2; Metabolic Disease; Sleeve Gastrectomy
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Placement (Experimental): The subjects in this arm will receive the Self-Forming Magnet (SFM) System that will be used to create a duodenal-ileal diversion. Following the diversion creation, a sleeve gastrectomy will also be performed.
  Interventions: Device: Self Forming Magnetic (SFM) Anastomosis System

INTERVENTIONS:
Device: Self Forming Magnetic (SFM) Anastomosis System — The SFM will be placed using an endoscope in the duodenum and laparoscopically into the ileum. A compression anastomosis will be created in each of the subjects and the diversion of enteral flow from the duodenum to ileum will create a metabolic effect that will induce weight loss and impact Type 2 Diabetes. Following the diversion being created, a gastric sleeve will be created according to standard technique.

SUMMARY:
Study will monitor weight loss and metabolic indicators for subjects in multi-center, single arm trial.

DETAILED DESCRIPTION:
Multi-Center, Open-label Pilot Study to Evaluate the Safety and Effectiveness of the GI Windows Single Neodymium Magnet Anastomosis Procedure When Used to Create a Duodenal-Ileal Diversion with a Sleeve Gastrectomy (SNAP-S) for Subjects with Obesity and Type 2 Diabetes Mellitus (T2DM)

ELIGIBILITY:
Inclusion Criteria:

* Age 19-65 years at screening
* Body mass index (BMI) ≥35 and ≤50
* T2DM diagnosis ≥6 months but < 10 years, with 1 or more oral diabetes medications, HbA1c ≥ 6.5% but < 10.0% at time of enrollment.
* HbA1c must be stable over a 3-month period.
* Weight stable over 3-month period
* Obesity-related comorbidities (hypertension, dyslipidemia, sleep apnea) must be well-controlled
* Agrees to refrain from any type of additional bariatric or reconstructive surgery that would affect body weight for a duration of 2 years
* If female, subject must commit to not becoming pregnant for 24 months and agree to use contraception during this period
* Able to understand and sign informed consent documents.

Exclusion Criteria:

* Known or suspected allergy to nickel or titanium or nitinol
* Type 1 diabetes or poorly controlled type 2 diabetes
* Use of injectable insulin
* Any documented conditions for which endoscopy would be contraindicated
* Contraindication to general anesthesia
* History of chronic gastrointestinal disease
* Congenial or acquired anomalies of the GI tract
* Any previous major surgery on the stomach, duodenum, hepatobiliary tree (excluding gallbladder), pancreas, or right colon.
* Uncontrolled hypertension
* Pre-existing severe comorbid cardio-respiratory disease
* History of chronic gastrointestinal disease
* Specific genetic or hormonal cause of obesity
* Recent tobacco/nicotine product cessation (within 3 months prior)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 12 months
  Weight loss measured as a percent of total body weight (TBW)

SECONDARY OUTCOMES:
Percent Responders | 12 months
  Percent responders; i.e. percent of subjects losing at least 10% TBW
Excess Weight Loss Measures | 12 months
  Excess weight loss (EWL)
Absolute Weight Loss Measures | 12 months
  Absolute weight loss
BMI - Weight Loss Measures | 12 months
  Change in BMI
Fasting Glucose | 12 months
  Mean change in fasting glucose
Hemoglobin A1c | 12 months
  Mean change in Hemoglobin A1c
Diabetes Remission and/or Improvements | 12 months
  Proportion of subjects experiencing diabetes remission and/or improvements
Diabetes Medication Dosage and Frequency Changes | 12 months
  Mean change in the dosage and frequency of diabetes medications from baseline
Serum Lipids | 12 months
  Mean change in serum lipids
Blood Pressure Changes | 12 months
  Mean percent change in systolic/diastolic blood pressure
Liver Changes using Fibroscan | 12 months
  Change in Controlled Attenuation Parameter (CAP) Scores from baseline
Nutritional Status | 12 months
  Nutritional Status: changes in pre-albumin levels
Albumin - Nutritional Status | 12 months
  Nutritional Status: changes in albumin levels

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No